CLINICAL TRIAL: NCT07384910
Title: Assessment of GARP Expression and Inflammatory Cytokines in Acute and Chronic Coronary Syndrome
Brief Title: Assessment of GARP Expression in Acute and Chronic Coronary Syndrome
Acronym: GARP-CS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Université Catholique de Louvain (Other)
Collaborators: Fonds National de la Recherche Scientifique (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: GARP-CS
Record Dates: First submitted 2026-01-26; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Atheroma; Heart
Keywords: Atheroma; Atherosclerosis; GARP; LRRC32
MeSH Terms: conditions — Coronary Artery Disease; Plaque, Atherosclerotic; Atherosclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Acute coronary syndrome (Experimental): This arm includes patients undergoing coronary angiography with a final diagnostic of acute coronary syndrome. The intervention administered is an arterial blood sample from the sheath at the beginning of the examination.
  Interventions: Biological: Arterial blood sample
- Chronic coronary syndrome (Experimental): This arm includes patients undergoing coronary angiography with a final diagnostic of chronic coronary syndrome. The intervention administered is an arterial blood sample from the sheath at the beginning of the examination.
  Interventions: Biological: Arterial blood sample
- Control (Experimental): This arm includes patients undergoing coronary angiography with a final diagnostic of non significant coronary disease. The intervention administered is an arterial blood sample from the sheath at the beginning of the examination.
  Interventions: Biological: Arterial blood sample

INTERVENTIONS:
Biological: Arterial blood sample — An arterial blood sample will be obtained at the beginning of the coronary angiography by using the arterial sheat in place.

SUMMARY:
The leading cause of death is cardiovascular diseases in occidental countries. Of those, atherosclerosis is the major contributor to this burden being notably responsible for strokes and myocardial infarctions. The genesis of atherosclerosis is linked to both lipid accumulation and inflammation in the vascular wall of major arteries. One of the major pathways of inflammation is the TGF-beta axis which is at least partially regulated by the GARP protein. It has been investigated mostly in cancer biology but data in cardiovascular disease is lacking. Thus, the investigators aim to characterize the contribution of this protein by investigating its expression in circulating blood cells from patients with an acute or chronic coronary syndrom. The main cells expressing the GARP protein are the platelets and the T regulating cells which will be the main focus.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years
* Able to give informed consent
* Undergoing coronary angiography.

Exclusion Criteria:

* Patients younger than 18 years
* Unable to give consent
* Pregnancy
* Dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Platelet GARP expression | Throughout the entire study, approximately during 2 years
  The platelet GARP expression profile will be assessed and compared between arms using flow cytometry.

SECONDARY OUTCOMES:
Inflammatory profile | Throughout the entire study, approximately during 2 years
  The inflammatory cytokines profile will be determined by multiplex and compared between arms.

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Beauloye, Medical Degree, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (1):
- Cliniques Universitaires Saint-Luc, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No